CLINICAL TRIAL: NCT04364178
Title: Viral Specific T-Lymphocytes by Cytokine Capture System (CCS) to Treat Infection With Adenovirus or Cytomegalovirus After Hematopoietic Cell Transplantation or Solid Organ Transplantation and in Patients With Compromised Immunity
Brief Title: Viral Specific T-Lymphocytes to Treat Adenovirus or CMV
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jessie L. Alexander (Other)
Responsible Party: Sponsor-Investigator, Jessie L. Alexander, Clinical Associate Professor of Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69251
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Adenovirus; Cytomegalovirus Infections
Keywords: Cytokine Capture System; Adenovirus; Cytomegalovirus; Hematopoietic Cell Transplant; Solid Organ Transplant; Immunocompromised; Inborn Error of Immunity
MeSH Terms: conditions — Adenoviridae Infections; Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Viral Specific T-Lymphocytes (Experimental): Peripheral blood mononuclear cells will be collected from the donor and loaded onto our Miltenyi Biotec CliniMACS Prodigy® or CliniMACS® Plus where they will be stimulated in vitro with viral-specific antigen(s). The cells are then immunomagnetically labeled with interferon gamma via the cytokine capture system. By this method, viral specific, gamma-secreting T cells, are captured in a closed, sterile system.
  Interventions: Biological: Adenovirus Specific T- Lymphocytes; Biological: Cytomegalovirus Specific T-Lymphocytes

INTERVENTIONS:
Biological: Adenovirus Specific T- Lymphocytes — Peripheral blood mononuclear cells will be collected from the donor and loaded onto our Miltenyi Biotec CliniMACS Prodigy® or CliniMACS® Plus where they will be stimulated in vitro with Adenovirus viral-specific antigen(s). The cells are then immunomagnetically labeled with interferon gamma via the cytokine capture system, captured and infused.
Biological: Cytomegalovirus Specific T-Lymphocytes — Peripheral blood mononuclear cells will be collected from the donor and loaded onto our Miltenyi Biotec CliniMACS Prodigy® or CliniMACS® Plus where they will be stimulated in vitro with Cytomegalovirus viral-specific antigen(s). The cells are then immunomagnetically labeled with interferon gamma via the cytokine capture system, captured and infused.

SUMMARY:
The primary purpose of this phase I/II study is to evaluate whether partially matched, ≥2/6 HLA-matched, viral specific T cells have efficacy against adenovirus and CMV in subjects who have previously received any type of allogeneic HCT or solid organ transplant (SOT), or have compromised immunity. Reconstitution of anti-viral immunity by donor-derived cytotoxic T lymphocytes has shown promise in preventing and treating infections with adenovirus and CMV. However, the weeks taken to prepare patient-specific products, and cost associated with products that may not be used limits their value. In this trial, we will evaluate viral specific T cells generated by gamma capture technology. Eligible patients will include HCT and/or SOT recipients, and/or patients with compromised immunity who have adenovirus or CMV infection or refractory viremia that is persistent despite standard therapy. Infusion of the cellular product will be assessed for safety and efficacy.

DETAILED DESCRIPTION:
If a subject shows a partial response, defined as a decrease in viral load of at least 50% from baseline or 50% improvement of clinical signs and symptoms, or no response, they are eligible to receive up to 4 additional cellular infusions from the same donor, at a minimum of 14-day intervals. If the same donor is no longer available, eligible, or appropriate, another donor may be considered for a maximum of 4 total cellular infusions at the discretion of the study PI and treating physician. A subject will not exceed a maximum of 5 total infusions from 2 donors.

Subjects are followed for 1 year post initial viral-specific T cell infusion. If subjects receive additional infusion(s), GvHD and adverse events will be followed for an additional 90 days from last infusion. Data may be abstracted from subjects' medical charts for an additional 1 year after most recent viral-specific T cell infusion.

ELIGIBILITY:
1. Patient, parent, or legal guardian must have given written informed consent, according to FDA guidelines. For patients ≥ 7 years of age who are developmentally able, assent or affirmation will be obtained, if feasible.
2. Male or female, 1 month through 60 years old, inclusive, at the time of informed consent.
3. Prior allogeneic hematopoietic stem cell transplant (bone marrow, peripheral blood stem cells, single or double cord blood), OR prior solid organ transplant (liver, kidney, lung and/or heart, intestinal, or multivisceral), OR diagnosis of primary immunodeficiency OR current/recent administration of immunosuppressive therapy for cancer or autoimmune disease.
4. Clinical status, at time of consent, amendable to tapering of steroids to less than 1 mg/kg/day prednisone (or equivalent) prior to cellular infusion.
5. Negative pregnancy test for females ≥10 years old or who have reached menarche, unless surgically sterilized.
6. Diagnosis of Adenovirus or CMV infection, persistent despite standard therapy.

   A. Adenovirus Infection or Disease:
   1. Active adenovirus infection: (i.e. gastroenteritis, pneumonia, hemorrhagic cystitis, hepatitis, pancreatitis, meningitis) defined as the demonstration of adenovirus by biopsy specimen from affected site(s) (by culture or histology), or the detection of adenovirus by culture, PCR or direct fluorescent antibody stain in fluid in the presence of worsening or persistent clinical or imaging findings despite at least 14 days of appropriate antiviral therapy (i.e. cidofovir, brincidofovir, or other available pharmacological agents) OR
   2. Refractory adenoviremia: defined as DNAemia >5000 copies/mL or <1 log decrease after at least 2 weeks of appropriate antiviral therapy (i.e. cidofovir, brincidofovir, or other available pharmacological agents) OR
   3. Intolerance of or contraindication to antiviral medications.

   B. CMV Infection or Disease:
   1. Active CMV infection: (i.e. pneumonia, meningitis, retinitis, hepatitis, hemorrhagic cystitis, and/or gastroenteritis) defined as the demonstration of CMV by biopsy specimen from affected site(s) (by culture or histology) or the detection of CMV by culture, PCR or direct fluorescent antibody stain in fluid in the presence of worsening or persistent clinical or imaging findings despite at least 14 days of appropriate antiviral therapy (i.e. Foscarnet, ganciclovir, cidofovir, or other available pharmacological agents) OR
   2. Refractory CMV viremia: defined as the continued presence of DNAemia, with ≥2,000 IU/mL or <1 log decrease after at least 14 days of appropriate antiviral therapy (i.e. Foscarnet, ganciclovir, cidofovir, or other available pharmacological agents) OR
   3. Intolerance of or contraindication to antiviral medications.
7. Donor Eligibility Criteria

   1. 12 years of age or older
   2. Able to understand and consent/assent to the procedure
   3. Required hemoglobin of 11g/dL

Exclusion Criteria:

1. Received ATG or Alemtuzumab within 28 days of viral-specific T cell infusion and a lack of evidence of T cell survival, defined by <10 CD3+ T cells/uL (in unique situations, plasmapheresis may be considered).
2. Active acute GVHD grades II-IV.
3. Active severe chronic GVHD.
4. Received donor lymphocyte infusion, with the exception of a fraction of an umbilical cord blood, within 21 days of viral-specific T cell infusion. Subjects receiving a fraction of an umbilical cord blood within 21 days of the viral-specific T cell infusion will not be excluded.
5. Active and uncontrolled relapse of malignancy.
6. Anticipated initiation of new lymphotoxic therapy within 4 weeks of viral-specific T cell infusion.
7. Patients who are pregnant or lactating.
8. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks to participation in the study, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study.
9. Donor Exclusion Criteria

   1. Patients who are pregnant
   2. Patients who are HIV positive
   3. Uncontrolled infection
   4. Deemed high risk due to pre-existing medical condition

Ages: 1 Month to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Grade III-IV Acute Graft versus host disease | Day 0 through 90 days after last cellular infusion
  The number of patients who develop Grade III-IV acute graft versus host disease (GVHD) attributed to the viral specific T cells.
CTCAE Grade 4/5 Adverse Events | Day 0 through 30 days from last cellular infusion
  The incidence of patients who develop CTCAE Grade 4/5 Adverse events

SECONDARY OUTCOMES:
6-month Survival (continuous) | First cellular infusion to 6 months post first cellular infusion
  Number of deaths that occurred from treatment
Viral load by Polymerase Chain Reaction (PCR) | Baseline through study completion, an average of 6 months
  The pace at which the viral load is undetectable in whole blood or plasma
Viral load from Respiratory Viral Panel (RVP) | Baseline through study completion, an average of 6 months
  The pace at which the viral load is undetectable from nasopharyngeal swab
Viral load from Bronchoalveolar lavage (BAL) | Baseline through study completion, an average of 6 months
  The pace at which the viral load is undetectable from bronchial washing
Viral load from Urine | Baseline through study completion, an average of 6 months
  The pace at which the viral load is undetectable from urine sample
Viral load from Stool | Baseline through study completion, an average of 6 months
  The pace at which the viral load is undetectable from stool sample
Viral load from fluid/tissue | Baseline through study completion, an average of 6 months
  The pace at which the viral load is undetectable from other fluid/tissue sample
Clinical response to viral specific infusion | Baseline through study completion, an average of 6 months as clinically indicated
  By imaging and symptomatology
Antiviral Agents | Day 0 through study completion, an average of 6 months
  The introduction of concomitant antiviral medication post infusion, if any
Immune Reconstitution | Baseline through study completion, an average of 6 months
  The pace of systemic immune reconstitution

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Alexander, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Jessie Alexander, Palo Alto, California
  - Lucile Packard Children's Hospital, Palo Alto, California

IPD SHARING:
Plan to Share IPD: No